CLINICAL TRIAL: NCT03000972
Title: PFN-A Intramedullary Nail and Intertrochanteric Hip Fracture. Augmentation of the Femoral Head Assessed by PET-CT (Positron Emission Tomography - Computed Tomography)- a Randomized Trial
Brief Title: PFN-A Augmentation for Intertrochanteric Femoral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PFNA
Record Dates: First submitted 2016-11-10; First posted 2016-12-22 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Intertrochanteric Fracture
Keywords: Augmentation; PET-CT; Positron Emission Tomography; Fluorine-18
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Nail (Active Comparator): Hip fracture surgery with a PFN-A Nail (Proximal Femoral Nail Augmentation).
  Interventions: Procedure: PFN-A Nail
- Augmented Nail (Experimental): Hip fracture surgery with a PFN-A Nail with Cement augmentation with TraumaCemV+
  Interventions: Procedure: Cement augmentation; Procedure: PFN-A Nail

INTERVENTIONS:
Procedure: Cement augmentation
  Arms: Augmented Nail
Procedure: PFN-A Nail

SUMMARY:
This study evaluates the potential negative effect of cement augmentation in the femoral head on viability of the head. Half of the participants will have the standard intramedullary nail (PFN-A; Proximal Femoral Nail Augmentation), while the other half will get the standard nail plus cement augmentation.

DETAILED DESCRIPTION:
Cement augmentation is believed to increase the bone implant interface and therefore decrease the risk of implant cut-out of the femoral head. The cement used in previous studies has produced heat and thermal necrosis on bone cells. The cement used in this study (TraumaCemV+) is manufactured specially for this implant and for the augmentation of this implant. TraumaCemV sets under low temperature (40 degrees Celsius) and we do not anticipate any heat necrosis. The volume effect of the cement could theoretically also damage the blood flow in the femoral head. There have been no negative effects in big series of patients operated with this technique.

The aim of this study is to quantify the viability of the femoral head with the use PET-CT (Positron Emission Tomography with simultaneous Computed Tomography) including a radioactive isotope (Fluorine-18) and the use of threedimensional computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Intertrochanteric Hip Fracture AO (Arbeitsgemeinschaft für Osteosynthesefragen) 31-A1 or AO 31-A2
* Healthy contralateral hip
* ASA (American Society of Anesthesiologists) Physical Status Class I or II

Exclusion Criteria:

* Dementia

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Viability of the femoral head as assessed by fluoride uptake using PET-CT | 4 months postoperatively
  The primary endpoint is the level of fluoride uptake (standardized uptake values: SUVs) representing bone metabolism. PET-CT enables us to quantify this tridimensionally.

SECONDARY OUTCOMES:
Viability of the femoral head as assessed by fluoride uptake using PET-CT | Within 1 week postoperatively
Viability of the femoral head as assessed by fluoride uptake using PET-CT | 1 year postoperatively
Harris Hip Score | 4 months
Harris Hip Score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Olof Wolf, MD PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No